CLINICAL TRIAL: NCT03192852
Title: Evaluation of Bleaching In-office With Violet LEd Light (405 nm): Randomized, Controlled Double Blind and Clinical Trial
Brief Title: Evaluation of Dental Bleaching In-office
Acronym: Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Professor of postgraduate program in Biophotonics Applied to Health Sciences, University of Nove de Julho, UNINOVE, São Paulo, Brazil, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2.034.518
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2018-07

CONDITIONS: Esthetics, Dental
Keywords: Tooth bleaching color; dental esthetic; Clinical Trial; Violet LED light; Violet LED; color; sensibility; dental aesthetic
MeSH Terms: interventions — tooth-bleaching agent, Opalescence; Gingivoplasty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: We will use a gel with no effect only in the fourth session of group 3 to match the number of sessions in relation to the other groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Violet LED (405 nm)+ gel placebo (Experimental): 20 patients will be submitted to dental bleaching involving the teeth 15-25 and 45 - 35 with Violet LED 405 nm (Bright Max Whitening, MMO, São Carlos, SP, Brazil) with gingival barrier + gel placebo
  Interventions: Other: dental bleaching
- Violet LED + CP 35% (Active Comparator): 20 patients will be submitted to dental bleaching involving the teeth 15-25 and 45 - 35 with carbamide peroxide 35% ( Whiteform - Fórmula & Ação, São Paulo, Brazil) actived with Violet LED 405 nm (Bright Max Whitening, MMO, São Carlos, SP, Brazil) with gingival barrier
  Interventions: Other: dental bleaching
- HP 35% (Active Comparator): 20 patients will be submitted to dental bleaching involving the teeth 15-25 and 45 - 35 with hydrogen peroxide 35% (Whiteness HP, FGM, Joinvile, SC, Brasil) and gingival barrier
  Interventions: Other: dental bleaching
- HP 35% + Violet LED + Gingivoplasty (Experimental): 20 patients will be submitted to dental bleaching involving the teeth 15-25 and 45 - 35 with Violet LED 405 nm (Bright Max Whitening, MMO, São Carlos, SP, Brazil) with gingival barrier split-mouth at first session. After 48 hours will be do Gingivoplasty.
  Interventions: Other: dental bleaching; Procedure: Gingivoplasty
- CP 35% (Active Comparator): 20 patients will be submitted to dental bleaching involving the teeth 15-25 and 45 - 35 with carbamide peroxide 35% ( Whiteform - Fórmula & Ação, São Paulo, Brazil)
  Interventions: Other: dental bleaching

INTERVENTIONS:
Other: dental bleaching — dental bleaching can be achieved with light, light+ peroxide carbamide gel, or only with peroxide carbamide gel
Procedure: Gingivoplasty — gengivoplasty will be realized to in illuminated tissue an no illuminated tissue to morphometrically evaluate the tissue
  Arms: HP 35% + Violet LED + Gingivoplasty

SUMMARY:
We aim to evaluate colorimetric changes after supervised whitening treatment, using Violet LED light associated or not with carbamide peroxide 35% gel. 80 will be divided into: Group 1 - Violet LED light, Group 2 Violet LED light + carbamide peroxide 35% gel, Group 3 -hydrogen peroxide 35% and Group 4 will be submitted to the gingivoplasty surgery procedure, for aesthetic desire, after whitening treatment with Violet LED light without gel. The colorimetric changes will be measured before, right after each whitening session in the end of the period of 3 months, through the Vitapan Classical (Vita) color scale, and by digital spectrophotometer. The sensibility degree will be measured by the Visual Analogue Scale (VAS) . The gum tissues Group 4, will be analyzed by histomorphometrically. Quality of life will be evaluated.

DETAILED DESCRIPTION:
This randomized, blind controlled trial has the objective of evaluate colorimetric changes after supervised whitening treatment, in-office, using Violet LED light of 405 nm associated or not to the use of carbamide peroxide 35% gel. Eighty patients, of which 20 with aesthetics desires to be submitted to gingivoplasty surgery, will be divided into four groups. Group 1 will receive whitening only with Violet LED light (405 nm). Group 2 will receive a whitening treatment combination of Violet LED light with carbamide peroxide 35% gel. Patients of Group 3 will receive a whitening treatment with hydrogen peroxide 35% and Group 4 will be submitted to the gingivoplasty surgery procedure, for aesthetic desire, after whitening treatment with Violet LED light (405 nm) without gel. The colorimetric changes will be measured before, right after each whitening session in the end of the period of 3 months, through the Vitapan Classical (Vita) color scale, and by digital spectrophotometer (SpectroShade™ Micro MHT Optic Research). The sensibility degree will be measured by the Visual Analogue Scale (VAS) in each session and in all groups. The gum tissues removed during the gingivoplasty in Group 4, will be histomorphometric analyzed to measure possible inflammatory gum changes by the Violet LED light (405 nm) irradiation. The degree of satisfaction of the patient and the life quality after aesthetic result achieved will be evaluated. The results will be presented by means and standard deviation. After checking the normality of the data, a one-way ANOVA will be performed. In case the data do not follow a normal distribution, it will be utilized the Kruskal-Wallis test and a value of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* negative medical history,
* Good systemic and oral health
* Patients with aesthetic complaint of discoloration of upper and lower teeth
* Patients with aesthetic desire for gingivoplasty, regardless of color in the baseline (Group 4), without the need for a prosthetic procedure and with sufficient gingiva inserted
* Color in the baseline higher than the A2 of the vita scale for groups 1, 2 and 3.

Exclusion Criteria:

* Patients with dentin hypersensitivity, incisal and occlusal wear or open cavities;
* Patients with pulp alterations;
* Carriers of dental anomalies;
* Patients with dental fractures who do not have restorations on the buccal surface of the teeth to be cleared;
* Patients who have had dental bleaching for less than 2 years;
* Holders of fixed appliances, orthopedic;
* Teeth pigmented by intrinsic factors;
* Smokers;
* Pregnant and Infants;
* Patients reporting adverse reactions to Hydrogen Peroxide;
* Patients who are taking ferrous sulfate medication;
* Patients who use chronic decorticosteroids, as well as volunteers who are taking analgesics or anti-inflammatories.
* Individual or removable prosthesis holders on the analyzed teeth will also be excluded or patients with endodontically treated teeth (Teeth 15-25 and 45-35).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Color Evaluation | baseline
  Color evaluation will be done before and after each bleaching session through the Vita Classical scale (VITA Zanhnfabrik, BadSӓckingrn, Germany) and SpectroShade ™ Micro MHT Optic Research by a previously trained and blind evaluator in the 4 groups
Color Evaluation | 3 months
  Color evaluation will be done 3 months after bleaching through the Vita Classical scale (VITA Zanhnfabrik, BadSӓckingrn, Germany) and SpectroShade ™ Micro MHT Optic Research by a previously trained and blind evaluator in the 4 groups

SECONDARY OUTCOMES:
Pain measured with Visual Analogue Scale (VAS) | baseline
  The pain will be evaluated through the Visual Analogue Scale (VAS) at each session before and after bleaching in the 4 groups.
Pain measured with Visual Analogue Scale (VAS) | 3 months
  The pain will be assessed through the Visual Analogue Scale (VAS) 3 months after the end of tooth whitening in the 4 groups.
Quality of life measured with Psychosocial Impact Questionnaire | baseline
  Quality of life will be assessed through the Psychosocial Impact of Dental Aesthetics Questionnaire validated for Brazil at the Federal University of São Paulo (UNIFESP)
Quality of life measured with Psychosocial Impact Questionnaire | 3 months
  Quality of life will be evaluated through the Psychosocial Impact Questionnaire of the Dental Internship validated for Brazil at the Federal University of São Paulo (UNIFESP) 3 months after the end of the bleaching.
Histomorphometric evaluation | baseline
  will be histomorphometric analyzed to measure possible inflammatory gum changes by the Violet LED light (405 nm) irradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Ana EC Santos, MS, Study Chair — University of Nove de Julho
Locations (1):
- University of Nove de Julho (UNINOVE), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
After completing the data search, it is published in indexed journals with high impact factor

REFERENCES:
- [Derived] Santos AECG, Bussadori SK, Pinto MM, Brugnera AJ, Zanin FAA, Silva T, Martinbianco ALC, Pantano Junior DA, Rodrigues MFSD, Artese HPC, Deana AM, Motta LJ, Horliana ACRT. Clinical evaluation of in-office tooth whitening with violet LED (405 nm): A double-blind randomized controlled clinical trial. Photodiagnosis Photodyn Ther. 2021 Sep;35:102385. doi: 10.1016/j.pdpdt.2021.102385. Epub 2021 Jun 9. PMID 34116249
- [Derived] Santos AECGD, Bussadori SK, Pinto MM, Pantano Junior DA, Brugnera A Jr, Zanin FAA, Rodrigues MFSD, Motta LJ, Horliana ACRT. Evaluation of in-office tooth whitening treatment with violet LED: protocol for a randomised controlled clinical trial. BMJ Open. 2018 Sep 4;8(9):e021414. doi: 10.1136/bmjopen-2017-021414. PMID 30181185